CLINICAL TRIAL: NCT02632279
Title: Tryptophan Depletion in Parkinson's Disease Patients Treated With Deep Brain Stimulation of the Subthalamic Nucleus: Effects on Mood and Motor Functions
Brief Title: Tryptophan Depletion in PD Patients Treated With STN DBS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: * Insufficient rates of participant accrual
  * Effects in opposite direction of hypothesis
  * Study was not feasible
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Netherlands Brain Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Tryptophan depletion in PD
Record Dates: First submitted 2015-11-26; First posted 2015-12-16 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Deep Brain Stimulation; Subthalamic nucleus; Tryptophan depletion; Serotonin
MeSH Terms: conditions — Parkinson Disease | interventions — Tryptophan; tryptophyltryptophan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRP depleted (Experimental): TRP depleted protein drink
  Interventions: Dietary Supplement: Tryptophan (TRP) depletion; Device: Stimulator ON; Device: Stimulator OFF
- Placebo (Placebo Comparator): Balanced protein drink (+1.21g of TRP)
  Interventions: Dietary Supplement: Placebo; Device: Stimulator ON; Device: Stimulator OFF

INTERVENTIONS:
Dietary Supplement: Tryptophan (TRP) depletion — TRP depletion will be accomplished by administering a TRP-low amino acid protein drink containing 100 g of gelatin powder. The protein mixture consists of 18 amino acids. According to Dutch law, TRP is considered a food supplement and is not registered as a medicine.
  Other Names: TRP depleted
  Arms: TRP depleted
Dietary Supplement: Placebo — The placebo treatment will consist of an identical amino acid protein drink containing 100 g of gelatin powder to which 1.21g TRP is added.
  Arms: Placebo
Device: Stimulator ON — Participants will be tested while their stimulator is turned ON
Device: Stimulator OFF — Participans will be tested while their stimulator is turned OFF

SUMMARY:
The purpose of this study is to assess the effect of tryptophan depletion on mood and behavior in Parkinson's disease (PD) patients treated with deep brain stimulation (DBS) of the subthalamic nucleus (STN). By doing this, the investigators hope to be able to identify risk factors for and mechanisms underlying psychiatric side effects of STN DBS. The study will be an intervention study with a placebo controlled, randomized cross-over design.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder characterized by motor symptoms such as tremor, rigidity and slowness of movement. In later stages of the disease, when pharmacological treatment becomes less efficient, deep brain stimulation (DBS) of the subthalamic nucleus (STN) becomes a treatment option. Although motor symptoms improve significantly by DBS, a number of operated patients experience severe side effects, mostly related to mood, cognition or behavior. These adverse effects are most likely mediated through the serotonin (5-HT) system. Additionally, a dysfunction of the 5-HT system is implied in the pathophysiology of PD. PD patients are therefore regarded as 'vulnerable' to experiencing mood, cognitive and emotional problems due to changes in 5-HT activity.

To elucidate whether STN DBS is indeed the trigger for psychiatric and cognitive problems to arise in the PD patient, the 5-HT levels in PD patients implanted with STN DBS will be manipulated. In order to do this, the investigators will make use of the tryptophan (TRP) depletion method, an established research paradigm. In TRP depletion, the brain is depleted of TRP, the precursor of 5-HT, which consequently leads to lowered 5-HT levels. In both the normal and 5-HT depleted condition, mood- and cognitive parameters of the PD patients both with the STN stimulation on (ON) and off (OFF) will be assessed.

The goal is to get more insight into the effects of STN DBS in PD patients with a 5-HT vulnerabililty and the effects on 5-HT related mood and cognitive behaviour. This way, possible risk factors for and mechanisms underlying psychiatric side effects of STN DBS can be identified. The study is an intervention study with a placebo controlled, randomized cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* subjects must be mentally competent
* subjects must have undergone STN DBS surgery for PD symptomatology

Exclusion Criteria:

* head injury
* stroke
* currentl malignancy or infection
* neurological disorders other than PD
* psychoactive medication: specifically antidepressants and antipsychotics ( a stable dose of benzodiazepines will be allowed)
* clinically relevant cognitive decline, operationalized as a MMSE score < 24
* current psychiatric syptomatology, operationalized as a Hamilton Depression scale score > 16 or a score >2 on one of the MDS-UPDRS section I, items 1-6

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Mood | There will be 6 measurements spread over 2 testing days with a wash-out period of min. 1 weak. baseline measure, 3.5 hours after intake of the amino acid mixture, and 5.5 hours after intake of the amino acid mixture
  as assessed through the Profile of Mood States

SECONDARY OUTCOMES:
Motor scores | There will be 6 measurements spread over 2 testing days with a wash-out period of min. 1 weak. baseline measure, 3.5 hours after intake of the amino-acid mixture, and 5.5 hours after intake of the amino-acid mixture
  as assessed through the MDS-UPDRS
Impulsivity | There will be 6 measurements spread over 2 testing days with a wash-out period of min. 1 weak. baseline measure, 3.5 hours after intake of the amino-acid mixture, and 5.5 hours after intake of the amino-acid mixture
  as assessed through a reaction time task
Emotional Responsiveness | There will be 4 measurements spread over 2 testing days with a wash-out period of min. 1 weak. baseline measure, 3.5 hours after intake of the amino-acid mixture
  as assessed through the emotional responsiveness task

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Temel, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands